CLINICAL TRIAL: NCT00130585
Title: The Relative Bioavailability of Folate From a Mixed Diet Compared to Synthetic Folic Acid Using a Stable Isotope Method
Brief Title: Bioavailability of Folate From a Mixed Diet Using a Stable Isotope Method
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wageningen Centre for Food Sciences (Other)
Collaborators: Wageningen University (Other)
Organization: Wageningen University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: A-007-RW
Record Dates: First submitted 2005-08-12; First posted 2005-08-15 (Estimated); Last update posted 2005-10-04 (Estimated); Status verified 2005-08

CONDITIONS: Folate Bioavailability; Healthy
Keywords: Folate; Bioavailability; Stable isotopes

INTERVENTIONS:
Behavioral: Controlled diet
Behavioral: folic acid supplement
Behavioral: 13C11-labelled folic acid supplement

SUMMARY:
The main objectives of this project are:

1. to determine the relative bioavailability of dietary folate from a total diet, compared with synthetic folic acid and
2. to determine the bioavailability with a higher precision than previous methods.

The hypothesis is that the bioavailability of dietary folate within a confidence interval of +/-20% can be estimated.

DETAILED DESCRIPTION:
Folate plays a role in the prevention of certain birth defects and possibly also in prevention of neurocognitive diseases, cancer and cardiovascular disease. The proportion of dietary folate that is absorbed and becomes available for metabolic processes in the body has been estimated between 30 and 98%, but an accurate figure is lacking. Since subjects generally differ a lot in their folate or homocysteine response upon a change in dietary folate intake, the between-person variability in these responses is high. Therefore, bioavailability estimates derived from these responses have large confidence intervals. With this trial the researchers want to determine folate bioavailability with a higher precision than previous trials. A good estimate of folate bioavailability from the general diet is necessary to construct reliable dietary reference intakes for folate.

ELIGIBILITY:
Inclusion Criteria:

* Serum B12 >118pmol/L;
* Serum creatinine <125micromol/L;
* Plasma total homocysteine <26micromol/L.

Exclusion Criteria:

* Cardiovascular disease, cancer, rheumatoid arthritis, epilepsy, gastro-intestinal disorders;
* Use of drugs interfering with folate metabolism;
* Use of B vitamins within the period three months prior to the study.
* Body Mass Index (BMI) > 30

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 75
Dates: Start 2005-05; Study Completion 2005-06

PRIMARY OUTCOMES:
Bioavailability based on change in labelled folate concentration in plasma;
Bioavailability based on change in folate concentration in plasma

SECONDARY OUTCOMES:
Bioavailability based on change in concentration in plasma homocysteine

CONTACTS AND LOCATIONS:
Overall Officials: Petra Verhoef, Dr., Principal Investigator — Wageningen Centre for Food Sciences; Martijn Katan, Professor, Principal Investigator — Wageningen University
Locations (1):
- Wageningen University, Wageningen, Netherlands